CLINICAL TRIAL: NCT06255990
Title: Clinical and Histological Study of a Novel Dermal Substitute, NovoSorb® BTM, Used in the Treatment of Full-thickness Skin Defects
Brief Title: Clinical and Histological Study of a Novel Dermal Substitute
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Zurich (Other); Kantonsspital Aarau (Other); Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00828
Record Dates: First submitted 2024-01-31; First posted 2024-02-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Skin Transplantation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Punch biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NovoSorb® BTM and STSG: Full thickness skin defect qualifying for coverage with the dermal substitute NovoSorb® BTM before transplantation with a split-thickness skin graft (STSG) according to clinical routine
  Interventions: Other: Standard of care
- STSG alone: Full thickness skin defect qualifying for coverage with split-thickness skin graft (STSG) alone according to clinical routine
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Standard of care

SUMMARY:
The goal of this observational study is to compare a novel dermal substitute to a the current standard procedure in the treatment of full thickness skin defects.

The main questions aim to answer are:

• Is the skin elasticity treated with the novel dermal substitute better than the skin elasticity treated with the current standard procedure Participants skin elasticity will be measured by Cutometer® MPA-580 assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1 to 75 years
* Full-thickness skin defect qualifying for coverage with the dermal substitute NovoSorb® BTM before transplantation with a STSG:

  * Acute cases: burn injury, soft tissue injury, skin necrosis after purpura fulminans or similar condition
  * Reconstructive cases (elective surgery): e.g. scar formation after burn injury, giant congenital nevus, defect after removal of skin tumor, skin defect due to other surgical procedures
* Documented medical treatment decision of covering the full-thickness skin defects with either the two-step BTM/STSG procedure or with STSG alone or by using both techniques on different wound areas
* Informed consent by patients/parents or other legal representative

Exclusion Criteria:

* Infected wounds needing surgical procedure other than a dermal template
* Patients with known underlying or concomitant medical conditions that may interfere with normal wound healing (e.g. immune deficiency, systemic skin disease, any kind of congenital defect of metabolism including diabetes)
* Previous enrolment of the patient into the current study
* Adolescent/Adult patients or in case of children their parents/legal representatives unable to comply with the study protocol
* Adolescent/Adult patients or in case of children their parents/legal representatives having insufficient knowledge of local language
* Pregnant or breast feeding females

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The project population will consist of children and adults that received surgical coverage of full-thickness skin defects either the two-step BTM/STSG procedure or with STSG alone under routine conditions.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Skin elasticity after 1year post-transplantation | 1 year post-transplantation
  Comparison of skin elasticity of treated skin versus adjacent normal skin

SECONDARY OUTCOMES:
Histological staining | within 1 year after skin transplantation
  Histological characterisation of epidermal and dermal components
Skin color assessment | within 1 year after skin transplantation
  Changes in skin color
Photographical assessment | within 1 year after skin transplantation
  Changes in graft-size
Change of quality of life within one year after skin transplantation | within 1 year after skin transplantation
  Quality of life assessed with standard EuroQoL questionnaire
Immunohistochemical analyses | 14-21 days after BTM transplantation
  Histological characterisation of mature BTM

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Böttcher, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (4):
- Switzerland (4):
  - Cantonal Hospital Aarau, Aarau, Canton of Aargau
  - University Children's Hospital Zurich, Zurich, Canton of Zurich
  - University Hospital Zurich, Zurich, Canton of Zurich
  - Cantonal Hospital Winterthur, Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No